CLINICAL TRIAL: NCT07117123
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Postoperative Pharyngeal Pain During Thyroid Surgery Under General Anesthesia
Brief Title: Transcutaneous Electrical Acupoint Stimulation on Postoperative Pharyngeal Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, XiaoLiang Wang, Chief Physician, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY20250624-13
Record Dates: First submitted 2025-07-20; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Sore Throat After Thyroid Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAS group (Experimental): If you are randomly assigned to the transcutaneous electrical acupoint stimulation (TEAS) group, after you enter the anesthesia preparation, the doctor will stick special electrodes on your wrist (Lieque point) and the inside of your ankle (Zhaohai point), and connect the electrical stimulation device (Han's Pain Treatment Device, Nanjing Jisheng Medical Technology Co., Ltd., which has been clinically used and provided by this project team). The current intensity will gradually increase from a small amount to the maximum level you can tolerate (starting from 1mA, not exceeding the maximum safety range of 10mA). The entire transcutaneous electrical acupoint stimulation lasts for 30 minutes. This electrical stimulation is non-traumatic and painless. Most people only feel slight numbness, swelling, and heat.
  Interventions: Device: Transcutaneous electrical acupoint stimulation
- Control group (Placebo Comparator): Electrodes were applied to the same acupoints (bilateral Lieque and Zhaohai points), but no electrical stimulation was performed. Other operations were consistent with those in the intervention group.
  Interventions: Other: No electrical stimulation

INTERVENTIONS:
Device: Transcutaneous electrical acupoint stimulation — The doctor will stick special electrodes on your wrist (Lieque point) and the inside of your ankle (Zhaohai point), and connect the electrical stimulation device (Han's Pain Treatment Device, Nanjing Jisheng Medical Technology Co., Ltd., which has been clinically used and provided by this project team). The current intensity will gradually increase from a small amount to the maximum level you can tolerate (starting from 1mA, not exceeding the maximum safety range of 10mA). The entire transcutaneous acupoint electrical stimulation lasts for 30 minutes. This electrical stimulation is non-traumatic and painless. Most people only feel slight numbness, swelling, and heat.
  Arms: TEAS group
Other: No electrical stimulation — The doctor will attach special electrodes to your wrist (Lieque point) and the inside of your ankle (Zhaohai point), and connect them to an electrical stimulation device (Han's pain treatment device, Nanjing Jisheng Medical Technology Co., Ltd., which has been clinically used and is provided by this project team). No electricity (i.e. no stimulation)
  Arms: Control group

SUMMARY:
Thyroid surgery is a common type of surgery in thyroid and breast surgery, mainly used to treat benign and malignant thyroid diseases. Despite the continuous progress in surgical techniques and anesthesia management, postoperative sore throat (POST) is still one of the most common adverse reactions in the perioperative period. It is reported that the incidence of POST in patients undergoing general anesthesia is about 15%-62%, while the incidence in the thyroid surgery population can be as high as 68%-80%. POST not only increases the patient's postoperative discomfort, but also may affect swallowing and language functions, prolong hospitalization time, reduce the quality of postoperative recovery, and increase medical costs. Therefore, effectively reducing the incidence and severity of POST is of great significance for improving the prognosis of patients after thyroid surgery.

The mechanism of postoperative sore throat after thyroid surgery is relatively complex, mainly involving two aspects. First, endotracheal intubation is a necessary operation for general anesthesia. The mechanical stimulation, improper airbag pressure, unreasonable catheter model selection, and rough intubation operation can all lead to pharyngeal mucosal damage, congestion, and edema, thereby causing acute POST. Secondly, thyroid surgery itself may also cause pharyngitis, such as traction and compression of the trachea, recurrent laryngeal nerve and pharyngeal soft tissue during surgery, excessive backward tilt of the head and neck during surgery, and local stimulation caused by recurrent laryngeal nerve function monitoring. The above factors work together to cause the incidence and severity of POST in thyroid surgery patients to be significantly higher than other types of surgery.

At present, measures to reduce POST mainly include reducing the inner diameter of the tracheal tube, controlling the airbag pressure, lubricating the tracheal tube, and using glucocorticoids or local anesthetics, but the effect is limited, and some interventions have the risk of drug side effects. In recent years, transcutaneous electrical acupoint stimulation (TEAS) as a non-invasive and non-traumatic intervention has shown good application prospects in relieving perioperative stress, reducing nausea and vomiting, and promoting gastrointestinal function recovery. Studies have shown that TEAS can effectively relieve a variety of postoperative discomfort symptoms, including laryngeal discomfort and pharyngitis, by regulating the autonomic nervous system, activating the endogenous analgesic system, and reducing the levels of inflammatory factors (such as IL-6 and TNF-α).

Among the many optional acupoints, Lieque (LU7) and Zhaohai (KI6) have been used in the treatment of throat diseases in ancient literature due to their status as "eight meridian intersection points". Modern studies have also confirmed that this acupoint combination has a clear effect on improving throat foreign body sensation, pharyngeal pain and hoarseness. However, there is currently no prospective randomized controlled study focusing on Lieque and Zhaohai acupoints combined with TEAS intervention for people with throat pain after thyroid surgery. Therefore, this study intends to use TEAS intervention on bilateral Lieque and Zhaohai acupoints to comprehensively observe the effect on the incidence and severity of throat pain after thyroid surgery, and evaluate its effect on postoperative nausea and vomiting, anxiety scores and hemodynamic indicators, aiming to provide new non-drug intervention strategies and evidence-based basis for the management of accelerated recovery after thyroid surgery (ERAS).

The goal of this clinical trial is to evaluate whether transcutaneous electrical acupoint stimulation (TEAS) can reduce postoperative sore throat (POST) and improve recovery quality in adult patients undergoing thyroid surgery under general anesthesia.

The main questions it aims to answer are:

Can TEAS at bilateral LU7 (Lieque) and KI6 (Zhaohai) acupoints reduce the incidence and severity of POST within 48 hours after thyroid surgery? Does TEAS influence postoperative nausea and vomiting, anxiety scores, and perioperative hemodynamic stability? Researchers will compare a TEAS group receiving active electrical stimulation at LU7 and KI6 with a control group receiving sham stimulation without current to see if TEAS results in improved postoperative comfort and faster recovery.

Participants will:

Be randomly assigned to TEAS or control group Undergo TEAS or sham stimulation for 30 minutes before induction of anesthesia Receive standard general anesthesia and thyroid surgery Be followed up for 48 hours postoperatively for sore throat assessment, discomfort scores, and related indicators

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing thyroid surgery under general anesthesia, including both open and endoscopic approaches
* Provision of written informed consent by the patient or a legally authorized representative

Exclusion Criteria:

* Failed tracheal intubation or requirement for emergency tracheotomy during surgery
* Requirement for reoperation due to postoperative complications such as bleeding or nerve injury
* Presence of severe cardiopulmonary disease (ASA physical status ≥ IV) or long-term use of corticosteroids
* Incomplete clinical data or inability to complete follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Sore Throat (POST) at 24 Hours After Extubation | 24 hours after extubation
  The percentage of patients who report a POST score >1 at 24 hours following thyroid surgery under general anesthesia.
  Scoring Criteria:
  0 = No sore throat at any time after surgery
  1. = Mild sore throat (pain only on swallowing)
  2. = Moderate sore throat (pain at rest and worsens with swallowing)
  3. = Severe sore throat (requires analgesics or affects eating) Definition of Event: POST score >1 is defined as a positive occurrence.

SECONDARY OUTCOMES:
Incidence and Severity of POST at 1, 6, and 48 Hours After Extubation | 1 hour, 6 hours, and 48 hours after extubation
Incidence of Hoarseness of Voice (HOV) at 1, 6, 24, and 48 Hours After Extubation | 1 hour, 6 hours, 24 hours, and 48 hours after extubation
Duration of POST | Perioperative/Periprocedural
  Time from onset to complete resolution of postoperative sore throat symptoms, as recorded by the patient and confirmed by the investigator.
Incidence of Postoperative Nausea and Vomiting | Within 48 hours after surgery
  PONV incidence is defined as the occurrence of at least one of the following within the first 48 hours after surgery:
  1. Clinically significant nausea - Nausea severity measured using the Numerical Rating Scale for Nausea (0 to 10 points), where 0 = "No nausea" and 10 = "Worst imaginable nausea." A score of ≥ 4 is considered clinically significant nausea, indicating moderate or greater severity and potentially requiring antiemetic treatment.
  2. Vomiting or retching episodes - Any expulsion of gastric contents (vomiting) or heaving without expulsion (retching). Recorded as count data (integer ≥ 0).
  3. Use of rescue antiemetic medication - Administration of any antiemetic drug for treatment of nausea or vomiting within the observation period.
  Scale information:
  1. Numerical Rating Scale for Nausea:
  2. Minimum score: 0
  3. Maximum score: 10 Higher scores indicate worse nausea severity